



STUDY NUMBER: CASE 2918

ClinicalTrials.gov #: NCT03957876

Protocol Date: 18 January 2021

<u>STUDY TITLE:</u> A Phase II Study of CPX-351 as a Novel Therapeutic Approach for Patients with Myelodysplastic Syndromes (MDS) after Hypomethylating Agent Failure

PRINCIPAL INVESTIGATOR: Sudipto Mukherjee, MD, MPH

Taussig Cancer Center, Cleveland Clinic

Tel: 216-444-0506

E-mail: mukhers2@ccf.org

STATISTICIAN: Brian Hobbs

STUDY COORDINATOR: Allison Unger

Case Comprehensive Cancer Center

SPONSOR: Case Comprehensive Cancer Center

<u>SUPPORT/FUNDING</u>: Jazz Pharmaceutical

SUPPLIED AGENT(S): CPX-351

<u>IND #:</u> 143227

# **SUMMARY OF CHANGES**

| <b>Protocol Date</b> | Section | Change |
|---|---|---|
| Protocol Version 5.0 | | |
| 01/18/2020 | 20 All Updated PI and contact information to Dr. Mukherjee throughout protocol | |
| | 6.4 | Clarified adverse event reporting requirements during follow-up period. |
| | | Protocol Version 4.0 |
| 06/01/2020 | 1/2020 4.1 Updated inclusion criteria to include MDS/MPN | |
| 06/01/2020 | 4.1 | Updated inclusion criteria for creatinine requirements |
| | Protocol Version 3.0 | |
| 11/13/2019 | 1.2 | Corrected dosing reconstitution from 5mg - 8.8mg/mL to 5mg - 2.2mg/mL |
| 11/13/2019 9.1 Corrected dosing reconstitution from 5mg - 8.8mg/mL to 2.2mg/mL | | |
| 11/13/2019 | Added language which will allow ECHO, EKG and Bone marrow biopsy and aspirate to be used for screening if completed within 28 days of C1D1 and prior to consent. | |
| Added footnote r, which will allow ECHO, EKG and Bone biopsy and aspirate if completed prior to consent and within 2 C1D1 to be used for screening. | | |
| | | Protocol Version 2.0 |
| 09/18/2019 | 11.2 | Updated requirements of ECHO at C1D1. |
| 09/18/2019 | 11.2 | Removed serum chemistry from follow-up visits. |
| 09/18/2019 | 8/2019 11.2 Updated requirements of vitals at induction and during consolid | |
| | | Updated remission bone marrow biopsy from D28 +/- 7 days to D35 +/- 10 days. |
| 09/18/2019 | 11.2 | Removed windows from follow-up and survival follow-up visits. |
| 09/30/2019 | SOC | Updated summary of changes table. |
| | | Protocol Version 1.0 |
| 03/27/2019 | 4.1 | Changed inclusion criteria from serum creatinine to creatinine clearance, and changed bilirubin inclusion criteria |
| 03/27/2019 | 4.2 | Added criteria to exclude all patients with AML and Wilsons disease |
| 03/27/2019 | 6.1 | Added information regarding premedication |
| 03/27/2019 | 6.3 | Added new EOT criteria for toxicities |
| 03/27/2019 | 6.3 | Added new EOS criteria. Table 2. |
| 03/27/2019 | 11.2 | Changed frequency of ECHO to D1 of every cycle |
| 03/27/2019 | 14.0 | Added toxicity monitoring plan |

# **Protocol Summary**

| Protocol Number/Title | CASE 2918: A Phase II Study of CPX-351 as a Novel<br>Therapeutic Approach for Patients with Myelodysplastic<br>Syndromes (MDS) after Hypomethylating Agent Failure |
|---|---|
| Study Phase | Phase II |
| Brief Background/Rationale | Epigenetic changes such as alterations in DNA methylation and histone modification play an important role in the pathophysiology of myelodysplastic syndromes (MDS). While hypomethylating agents (HMAs) such as azacitidine and decitabine have become the standard of care for patients with higher-risk MDS, they have limited efficacy. Response rates range from 20-40% and last a median of 9-10 months. Complete remissions are rare and the majority (50-70%) of patients remains resistant/refractory to these drugs. The poor success of HMAs is due, in part, to the limited understanding of mechanisms that underlie resistance. Given the poor survival of patients who fail HMAs, novel agents that overcome HMAs failure are desperately needed. Despite several novel compounds that have been investigated at the time of HMA failure, no therapy has proven to show overall survival (OS) compared to conventional care. This in part is due to the lack of our understanding into the mechanisms of resistance to HMA and the failure of accurately risk stratifying patients in this setting. We have previously shown that IPSS, IPSS-R and other commonly used MDS prognostic models, (e.g., the World, Health, Organization, (WHO), classification based. |
| | World Health Organization (WHO) classification-based Prognostic Scoring System (WPSS), and the MD Anderson Prognostic Scoring System (MDAPSS) have limited predictive power in the HMA failure setting 1-4. We therefore developed and validated a new model to predict outcome of patients after hypomethylating agent failure (HMAF) that includes 6 clinical variables: age, performance status, complex cytogenetics (≥4 abnormalities), marrow blast percentage >20%, platelet count, and red cell transfusion dependency 4. This model separates patients into two risk categories: lower-risk, with a median OS of 11.0 months (95% CI 8.8-13.6); and higher-risk disease, with median OS of 4.5 months (95% CI 3.9-5.3) 4. The model |

| | was subsequently validated in an independent cohort of 223 MDS patients derived from the Groupe Francophone des Myélodysplasies (GFM) database and in a phase III randomized clinical trial. Thus, risk stratifying MDS patients by the new model at the time of HMA failure may open new opportunity for drug approvals in this setting 5-6. Identifying novel drugs that can improve the outcome of MDS patients after HMA failure remains an unmet need. |
|---|---|
| | Evaluate the efficacy of CPX-351 as measured by overall response rate (ORR), i.e. by IWG 2006 criteria for MDS patients after Hypomethylating agent failure. |
| Primary Objective | Endpoint and time frame: Overall response rate (ORR), i.e. by IWG 2006 criteria for MDS and patients at end of induction (C1D35 +/-10). |
| | • To determine the time to response (TTR) associated with CPX-351 in patients with MDS |
| | Endpoint and time frame: TTR associated with CPX-351 in patient with MDS at the end of induction (C1D35 +/-10). |
| | • To evaluate the duration of response (DOR) in patients achieving a response |
| Secondary Objective(s) | Endpoint and time frame: DOR in patients achieving a response at the time of response (C1D35 +/-10) and up to 1 year after the end of treatment. |
| | • To evaluate the event-free survival (EFS) and the overa survival (OS) probability of all patients enrolled in this trial. |
| | Endpoint and time frame: EFS and OS probability of all patients enrolled in this trial at end of induction (C1D35 +/-10) and up to 1 year after the end of treatment. |
| Estimated Study Duration | Estimated date first subject enrolled: March, 2019 Estimated date last subject enrolled: March, 2020 |
| Duration of Participation | Patient participation is expected to average 6 to 12 months |
| Sample Size | 25 patients |

CASE 2918 Protocol Version 5.0 18 January 2021

| Disease sites/Conditions | Myelodysplastic Syndrome (MDS) |
|---|---|
| | • CPX-351 44mg/m <sup>2</sup> (daunorubicin 44 mg/m <sup>2</sup> and cytarabine 100 mg/m <sup>2</sup> ), IV days 1, 3, and 5 during the induction phase. |
| Interventions | • CPX-351 15.4mg/m <sup>2</sup> (daunorubicin 15.4 mg/m <sup>2</sup> and cytarabine 35 mg/m <sup>2</sup> ), IV every 28 days for up to 4 cycles during the consolidation phase for patients achieving a response. |

# **Abbreviations**

| AE | Adverse Event |
|---|---|
| ALL | Acute Lymphoblastic Leukemia |
| ALT | Alanine Aminotransferase |
| AML | Acute Myeloid Leukemia |
| AML-MRC | Acute Myeloid Leukemia with Myelodysplasia Related Changes |
| ANC | Absolute Neutrophil Count |
| AST | Aspartate Aminotransferase |
| AZA | Azacitidine |
| BSA | Body Surface Area |
| BUN | Blood Urea Nitrogen |
| CCCC | Case Comprehensive Cancer Center |
| CCF | Cleveland Clinic Foundation |
| CI | Confidence Intervals |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CR | Complete remission |
| CRi | Complete remission with incomplete count recovery |
| CRF | Case Report Form |
| DAC | Decitabine |
| DCRU | Dahm's Clinical Research Unit |
| DLT | Dose Limiting Toxicity |
| DOR | Duration of response |
| DSMP | Data Safety Monitoring Plan |
| DSTC | Data Safety and Toxicity Committee |
| ECOG | Eastern Cooperative Oncology Group |
| EFS | Event free survival |
| EOS | End of Study |
| EOT | End of Treatment |
| FDA | Food and Drug Administration |
| FU | Follow-up |
| GCP | Good Clinical Practice |
| G-CSF | Granulocyte-colony stimulating factor |
| GM-CSF | Granulocyte-macrophage colony-stimulating factor |
| GFM | Groupe Francophone des Myélodysplasies |
| Hgb | Hemoglobin |
| HI | Hematologic Improvement |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HMA | Hypomethylating agent |
| HMAF | Hypomethylating agent failure |
| HR | Hazard Ratio |
| HSCT | Hematopoietic stem cell transplant |
| HU | Hydrea |

CASE 2918 Protocol Version 5.0 18 January 2021

| ICF | Informed Consent Form |
|---|---|
| ICH | International Conference on Harmonization |
| IEC | Institutional Ethics Committee |
| IRB | Institutional Review Board |
| IWG | International Working Group |
| LLN | Lower Limit of Normal |
| MDAPSS | MD Anderson Prognostic Scoring System |
| MDS | Myelodysplastic Syndrome |
| MPN | Myeloproliferative Neoplasm |
| ORR | Overall Response Rate |
| OS | Overall survival |
| PD | Progressive Disease |
| PI | Principle Investigator |
| PR | Partial remission |
| PRMC | Protocol Review and Monitoring Committee |
| SAE | Serious Adverse Event |
| SD | Stable Disease |
| SOC | Standard of Care |
| tAML | Therapy Related Acute Myeloid Leukemia |
| TLS | Tumor lysis syndrome |
| TTR | Time to response |
| UH | University Hospitals |
| ULN | Upper Limit of Normal |
| WHO | World Health Organization |
| WPSS | World Health Organization Classification-Based Prognosis |
| | Scoring System |

#### TABLE OF CONTENTS

## 1.0 INTRODUCTION

- 1.1 Background of Study Disease
- 1.2 Name/description of CPX-351
- 1.3 Rationale

## 2.0 OBJECTIVES

- 2.1 Primary Objective
- 2.2 Secondary Objective(s)

## 3.0 STUDY DESIGN

- 3.1 Study design
- 3.2 Number of Subjects
- 3.3 Replacement of Subjects
- 3.4 Expected Duration of Treatment and Subject Participation

## 4.0 SUBJECT SELECTION

- 4.1 Inclusion Criteria
- 4.2 Exclusion Criteria
- 4.3 Inclusion of Women and Minorities

## 5.0 REGISTRATION

## 6.0 TREATMENT PLAN

- 6.1 Treatment Regimen Overview
- 6.2 Phase I Dose Escalation
- 6.3 Definition of Dose Limiting Toxicity
- 6.4 General Concomitant Medications and Supportive Care Guidelines
- 6.5 Criteria for Removal from Study
- 6.6 Duration of Follow-Up

## 7.0 DOSE DELAYS / DOSE MODIFICATIONS

## 8.0 ADVERSE EVENTS AND POTENTIAL RISKS

- 8.1 Agent Adverse events
- 8.2 Definitions
- 8.3 Serious Adverse Event Report Form
- 8.4 Reporting Procedures for Serious Adverse Event
- 8.5 Serious Adverse Events and OnCore<sup>TM</sup>
- 8.6 Data Safety Toxicity Committee
- 8.7 Data and Safety Monitoring Plan

## 9.0 PHARMACEUTICAL INFORMATION

- 9.1 Investigational Agent(s)
- 9.2 Commercial Agent(s)

**CASE 2918** 

Protocol Version 5.0

18 January 2021

## 10.0 EXPLORATORY/CORRELATIVE

## 11.0 STUDY PARAMETERS AND CALENDAR

- 11.1 Study Parameters
- 11.2 Calendar

## 12.0 MEASUREMENT OF EFFECT

## 13.0 RECORDS TO BE KEPT/REGULATORY CONSIDERATIONS

- 13.1 Data Reporting
- 13.2 Regulatory Considerations

## 14.0 STATISTICAL CONSIDERATIONS

## **REFERENCES**

## **APPENDICES**

## **APPENDIX I:**

ECOG / Karnofsky Performance Status Criteria

## APPENDIX II:

STUDY DESIGN TIME POINT DEFINITIONS

## APPENDIX III:

RESPONSE CRITERIA FOR CONSOLIDATION PERIOD

## **APPENDIX IV:**

STUDY DESIGN TIME POINT DEFINITIONS

## APPENDIX V:

POST-HMA FAILURE MODEL

## 1.0 Introduction

## 1.1 Background of Study Disease

Epigenetic changes such as alterations in DNA methylation and histone modification play an important role in the pathophysiology of myelodysplastic syndromes (MDS). While hypomethylating agents (HMAs) such as azacitidine and decitabine have become the standard of care for patients with higher-risk MDS, they have limited efficacy. Response rates range from 20-40% and last a median of 9-10 months. Complete remissions are rare and the majority (50-70%) of patients remains resistant/refractory to these drugs. The poor success of HMAs is due, in part, to the limited understanding of mechanisms that underlie resistance. Given the poor survival of patients who fail HMAs, novel agents that overcome HMAs failure are desperately needed. Despite several novel compounds that have been investigated at the time of HMA failure, no therapy has proven to show overall survival (OS) compared to conventional care. This in part is due to the lack of our understanding into the mechanisms of resistance to HMA and the failure of accurately risk stratifying patients in this setting.

We have previously shown that IPSS, IPSS-R and other commonly used MDS prognostic models, (e.g., the World Health Organization (WHO) classification-based Prognostic Scoring System (WPSS), and the MD Anderson Prognostic Scoring System (MDAPSS) have limited predictive power in the HMA failure setting <sup>1-4</sup>. We therefore developed and validated a new model to predict outcome of patients after hypomethylating agent failure (HMAF) that includes 6 clinical variables: age, performance status, complex cytogenetics (≥4 abnormalities), marrow blast percentage >20%, platelet count, and red cell transfusion dependency <sup>4</sup>. This model separates patients into two risk categories: lower-risk, with a median OS of 11.0 months (95% CI 8.8-13.6); and higher-risk disease, with median OS of 4.5 months (95% CI 3.9-5.3) <sup>4</sup>. The model was subsequently validated in an independent cohort of 223 MDS patients derived from the Groupe Francophone des Myélodysplasies (GFM) database and in a phase III randomized clinical trial. Thus, risk stratifying MDS patients by the new model at the time of HMA failure may open new opportunity for drug approvals in this setting <sup>5, 6</sup>.

CASE 2918 Protocol Version 5.0 Identifying novel drugs that can improve the outcome of MDS after HMA failure remains an unmet need.

## 1.2 Name and Description of Investigational Agent CPX-351

#### 1.2.1 Preclinical Data

CPX-351 is a liposomal formulation of a fixed combination of the antineoplastic drugs cytarabine and daunorubicin. These two drugs are present inside the liposome in a 5:1 molar ratio. The liposome membrane is composed of distearoylphosphatidylcholine, distearoylphosphatidylglycerol and cholesterol in a 7:2:1 molar ratio. These liposomes have a nominal diameter of approximately 100nm and are suspended in sucrose. Sterilization is achieved by filtration through a 0.22 µm filter.

CPX-351 is provided as a sterile, pyrogen-free lyophilized formulation in 50 mL glass, single-use vials. Each vial contains 100mg/m<sup>2</sup> of CPX-351 where each vial contains 100 mg cytarabine and 44 mg daunorubicin base in liposomes. The lyophilized cake is reconstituted with sterile water for injection to obtain a homogeneous dispersion at 5 mg-2.2mg/mL (cytarabine-daunorubicin).

The pre-clinical pharmacology and toxicology are summarized in the Investigator's Brochure for CPX-351.

#### 1.2.2 Clinical Data

## Phase I study of CPX-351

In a phase 1 dose-escalation trial, CPX-351 induction was administered on days 1, 3, and 5 by 90-minute infusion to 48 relapsed or refractory patients with acute myeloid leukemia (AML) or high-risk myelodysplasia. Doses started at 3 mg/m² with dose doublings in single-patient cohorts until a pharmacodynamic effect (treatment-related adverse events or reduction in bone marrow cellularity or blast count) was observed, followed by 33% escalations in three patient cohorts until dose-limiting toxicity (DLT) occurred. The maximum-tolerated dose was 101 mg/m². DLTs consisted of hypertensive crisis, congestive heart failure, and prolonged cytopenias. Identified adverse events were similar with cytarabine and daunorubicin treatment. Response occurred at doses as low as 32 mg/m². Of 43 patients with AML, nine had complete response (CR) and one had CR

with incomplete platelet recovery; of patients with acute lymphoblastic leukemia (ALL), one of three had CR. Eight CRs were achieved among the 31 patients with prior cytarabine and daunorubicin treatment. CR in AML occurred in 5 of 26 patient's age  $\geq$  60 years and in 5 of 17 patients younger than 60 years of age. Median half-life was 31.1 hours (cytarabine) and 21.9 hours (daunorubicin), with both drugs and their metabolites detectable  $\geq$  7 days after the last dose. The targeted 5:1 molar ratio was maintained at all dose levels for up to 24 hours<sup>7</sup>.

## Phase II study of CPX-351

A randomized, multicenter, open-label, phase 2 trial was conducted to evaluate the efficacy and safety of CPX-351 compared with investigators' choice of first salvage treatment in adult patients with first relapse AML. The primary endpoint of the study was 1-year overall survival (OS), and Kaplan-Meier analysis did not show a significant difference between the two treatment groups (HR, 0.75; P = 0.33). Survival at 1-year was 36% and 27% (P = 0.33) for CPX-351 and salvage treatment arms, respectively. Patients were stratified at baseline according to the European Prognostic Index (EPI), and results showed that CPX-351-treated patients with the EPI-defined poor-risk strata demonstrated higher response rates (39.3% CPX-351 versus 27.6% salvage arm) and improvements in event-free survival (EFS) (HR, 0.63; P = 0.8) and OS (HR, 0.55; P = 0.22). The overall rates of grade 5 AEs were similar between the CPX-351 (23.5%) and salvage treatment arms (20.5%)8.

## Phase III study of CPX-351

A phase 3, randomized, multicenter, open-label study evaluated the efficacy and safety of CPX-351 compared with conventional 7 + 3 (cytarabine for 7 days plus daunorubicin for 3 days) regimen in adult patients (60 to 75 years) with newly-diagnosed therapy-related Acute Myeloid Leukemia (tAML) or Acute Myeloid Leukemia with Myelodysplasia related changes (AML-MRC). The primary efficacy endpoint was overall survival (OS). The results showed OS was significantly greater in the CPX-351 group compared with the 7 + 3 group. The median OS was 9.56 months with CPX-351 and 5.95 months with 7 + 3 (Hazard Ratio [HR] 0.69; P = 0.005). Grade 3-5 non-hematologic CASE 2918

adverse events (AEs) occurring  $\geq$  5% were similar between the two groups, except pneumonia (20% vs 15%) and bacteremia (10% vs 2%) were numerically higher in the CPX-351 compared with 7 + 3 groups, respectively. Also, median time to recovery of absolute neutrophil count (ANC)  $\geq$  500/ $\mu$ L and platelets  $\geq$  50,000/ $\mu$ L were longer in the CPX-351 group than 7 + 3 group<sup>9</sup>.

#### 1.4 Rationale

Treatment options are limited for patients diagnosed with MDS at the time of HMA failure. Although the outcome remains poor, hematopoietic stem cell transplant (HSCT) may prolong survival for a subset of patients<sup>10</sup>. However, achievement of CR prior to transplant is important for improved outcomes<sup>10</sup>. Treatment with 7+3 chemotherapy regimen has been used, resulting in a response rate of approximately 30% in this patient population. Especially, in patients who progress to AML<sup>11</sup>. Transplant remains an important option for these patients who can tolerate chemotherapy.

CPX-351 has shown better overall response rate and improved overall survival in patients with AML with underlying MDS changes compared to 7+3 suggesting that CPX-351 can be used in this patient population. Thus, we hypothesize that treating MDS patients, who failed or are intolerant to their initial treatment with HMA's, with CPX-351 will overcome HMA resistance and sensitize the MDS cells to this treatment.

## 2.0 Study Objectives

## 2.1 Primary Objective

• Evaluate the efficacy of CPX-351 as measured by overall response rate (ORR), i.e. by IWG 2006 criteria for MDS patients after Hypomethylating agent failure.

## 2.2 Secondary Objective(s)

- To determine the time to response (TTR) associated with CPX-351 in patients with MDS.
- To evaluate the duration of response (DOR)

• To evaluate the event-free survival (EFS) and the overall survival (OS) probability of all patients enrolled in this trial.

## 3.0 Study Design

## 3.1 Overview of Study Design

This is a phase II study of single agent CPX-351 administered at the standard FDA approved dose of 44 mg/m<sup>2</sup> (daunorubicin 44 mg/m<sup>2</sup> and cytarabine 100 mg/m<sup>2</sup>) intravenously on days 1, 3, 5 of the induction cycle. If patients achieve complete remission (CR), complete remission with incomplete count recovery (CRi) or partial remission (PR) (section 12.0, Table 2) they will be eligible to continue on to consolidation therapy, which will consist of CPX-351 at a dose of 15.4 mg/m<sup>2</sup> (daunorubicin 15.4 mg/m<sup>2</sup> and cytarabine 35 mg/m<sup>2</sup>) every 28 days Patients can receive up to 4 cycles of consolidation therapy.

## 3.2 Number of Subjects

Approximately 25 patients will be enrolled in this trial.

## 3.3 Replacement of Subjects

Patients who receive any doses of CPX-531 will be not be replaced. Patient's slots will only be replaced if they are discontinued from the study prior to dosing with CPX-351. Missed doses of CPX-351 will be re-administered at the discretion of the treating physician.

## 3.4 Expected Duration of Treatment and Subject Participation

Enrollment to this study is estimated to occur over three years. Upon signing consent, patients will undergo screening to determine if the patient meets all inclusion and exclusion criteria, as outlined in section 4.1 and 4.2. Following screening, all eligible patients will be enrolled and begin induction therapy which will occur over a 35 day cycle and/or at count recovery with CPX-351 dosing on days 1, 3 and 5.

CASE 2918 Protocol Version 5.0 18 January 2021 Patients who achieve a response (section 12.0, Table 2) may proceed with the consolidation phase of the trial with CPX-351 dosing on days 1 and 3 of every 28 days. Patients can receive up to 4 cycles of consolidation. Treatment will continue during the duration of the study unless patients exhibit evidence of treatment failure, disease progression, experience an unacceptable toxicity, or the investigator determines that discontinuation of treatment is in the best interest of the patient. Patients will be treated with CPX-351 based on a calculation determined from the patient's body surface area (BSA). BSA will be calculated before each day of dosing and will be based on the patient's height (measured at baseline) and weight (measured each visit).

## 4.0 Subject Selection

## 4.1 Inclusion Criteria

Each patient must meet all of the following inclusion criteria to be eligible for enrollment:

- 1. Patients must be  $\geq$  18 years of age
- 2. Patients must give voluntary written consent before performance of any study related procedures not part of standard medical care
- 3. Diagnosis of MDS or MDS/MPN according to 2016 WHO criteria<sup>12</sup>
- 4. Primary therapy failure with either hypomethylating agents (decitabine or azacitidine) defined as:
  - Progression (according to 2006 IWG criteria)<sup>13</sup> after initiation of azacitidine or decitabine treatment; or
  - Failure to achieve complete or partial response or hematological improvement (according to 2006 IWG)<sup>13</sup> after at least 4-6 cycles (4-weeks cycle) of azacitidine or decitabine; or
  - Relapse after initial complete or partial response or hematological improvement (according to 2006 IWG criteria)<sup>13</sup> observed after at least 4 cycles of azacitidine or decitabine.
- 5. Eastern Cooperative Oncology Group (ECOG) Performance Status < 2
- 6. Subjects must have normal organ and marrow function defined as:
  - If total bilirubin ≤ 2x upper limit of normal (≤ 3 x ULN if considered to be due to leukemic involvement or Gilbert's syndrome) at the discretion of the treating physician following discussion with PI) Patients with a bilirubin level of >3 mg/dL will be excluded

- Calculated creatinine clearance value of ≥ 30ml/min AND a serum creatinine ≤ 1.5mg/dL
- LVEF ≥ 50%

## 7. Female patients who:

- Are postmenopausal for at least 1 year before the screening visit, OR
- Are surgically sterile, OR
- Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose

## 8. Male patients who:

- Are surgically sterile, OR
- Agree to practice true abstinence from heterosexual contact or agree to use effective contraception without interruption during the study therapy and 90 days after the last dose

#### 4.2 Exclusion Criteria

The presence of any of the following will exclude a subject from study enrollment.

- 1. Prior treatment with CPX-351, or known hypersensitivity to CPX-351 or its components.
- 2. Prior treatment with intensive chemotherapy.
- 3. Patients with confirmed Wilson's disease will be excluded.
- 4. Diagnosis of acute myeloid leukemia (AML)
- 5. Any serious medical condition, laboratory abnormality, or psychiatric illness that, in the view of the treating physician, would place the participant at an unacceptable risk if he or she were to participate in the study or would prevent that person from giving informed consent.
- 6. Any active malignancy (unrelated, non-hematological malignancy) diagnosed within the past 6 months of starting the study drug (other than curatively treated carcinoma-in-situ of the cervix or non-melanoma skin cancer).
- 7. Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
- 8. Known history of HIV or active hepatitis B or C.
- 9. Active Wilsons disease
- 10. Major surgery within 2 weeks prior to study enrollment.

## 11. Pregnant or lactating females

12. Male and female patients who are fertile who do not agree to use an effective barrier methods of birth control (i.e. abstinence or 2 forms of contraception) to avoid pregnancy while receiving study treatment.

## 4.3 Inclusion of Women and Minorities

Men, women and members of all races and ethnic groups are eligible for this trial.

## 5.0 Registration

All subjects who have been consented are to be registered in the OnCore<sup>TM</sup> Database. For those subjects who are consented, but not enrolled, the reason for exclusion must be recorded.

All subjects will be registered through Cleveland Clinic and will be provided a study number by contacting the study coordinator listed on the cover page.

#### 6.0 Treatment Plan

# 6.1 Treatment Regimen Overview Consent and Screening

Upon signing consent, patients will begin the screening phase. The screening period begins the day the patient signs consent and can take place over a 28 day period leading up to dosing on day 1 (D1). During the screening period patients will be assessed to determine if they meet eligibility for this study per the inclusion and exclusion criteria as outlined in sections 4.1 and 4.2. Once the patient is deemed eligible they will be stratified into two arms based on the post-HMA failure model (Appendix V).

## Stratification

Prior to beginning treatment, all eligible patients will be stratified into low vs. high risk based on the post-HMA failure model (Appendix V)<sup>4</sup>. Seven patients will be enrolled into the low risk arm and seven patients will be enrolled into the high risk arm. Once 14 patients, across both arms, have been enrolled and evaluated for a response (D35 +/- 10 days bone marrow), an interim analysis will be conducted to determine benefit in

each arm. The arm with the greatest response will then enroll an additional 11 patients, for a total of 18 patients in that arm. Overall, this study will enroll 25 patients.

## Induction

The induction phase is defined as the time between the first day (D1) of study drug to day 35 and/or count recovery. During the induction phase of the study, all patients will be treated with the FDA approved standard dose of CPX-351 at 44mg/m² (daunorubicin 44 mg/m² and cytarabine 100 mg/m²) on days 1, 3, and 5. Study drug will be administered per the study calendar (section 11.2) unless patient exhibits any EOT criteria. Premedication with anti-emetics is recommended prior to treatment with CPX-351. No re-induction will be allowed and no day 14 bone marrow biopsy is required. A bone marrow biopsy and aspirate will be obtained on day 35 +/-10 days to confirm response. If no evidence of blasts > 5%, G-CSF will be allowed to improve counts at the discretion of the treating physician. Following the bone marrow, patients who meet the response criteria per section 12.0 can then continue onto the consolidation phase of this study.

## Consolidation

The consolidation phase is defined as C2D1 to C5D28 or once the patients meet EOT criteria (section 6.3, Table 1). Only patients with a documented response (CR, CRi, or PR) from the D35 (+/-10 days) bone marrow are eligible for consolidation therapy. Prior to the first cycle of consolidation therapy the patients must have a PS of 0-2. During the consolidation phase, CPX-351 must be given no earlier than 35 days after the start of induction and no later than 75 days after the start of induction. For all subsequent cycles, there must be at least 35 days between the start of each cycle. Patients must have recovered to ANC >500/  $\mu$ L and platelets >50,000/ $\mu$ L to be eligible for any consolidation therapy.

During the consolidation phase, CPX-351 will be given at 15.4 mg/m<sup>2</sup> (daunorubicin 15.4 mg/m<sup>2</sup> and cytarabine 35 mg/m<sup>2</sup>) on days 1 and 3 of each 28 day cycle. Consolidation therapy can be continued up to 4 cycles in the absences of toxicities or reasons that require discontinuation and/or any EOT criteria (section 6.3, Table 1).

CASE 2918 Protocol Version 5.0 18 January 2021 Premedication with anti-emetics is recommended prior to treatment with CPX-351. No other chemotherapy consolidation treatment is permitted. Only HSCT (hematopoietic

stem cell transplant) is permitted in place of, or following, chemotherapy consolidation.

Delays in administrating consolidation cycles will be allowed at the discretion of the

treating physician and after discussion with the PI.

**End of Treatment and Follow-up** 

At the point in which the patient completes therapy per protocol or meets any

EOT criteria (section 6.3, Table 1), the patient will enter into the follow-up period. The

patient will be followed for survival for 1 year and/or until death, whichever occurs first.

During the first 6 months of follow-up the patient will be seen in clinic as standard of

care (SOC) every 30 days, per the study calendar (section 11.2). End of study (EOS) is

defined as the time the patient completes 1 year of follow, withdraws consent and/or

patient's death, whichever occurs first.

6.1.1 Name of **Investigational Agent** 

CPX-351

6.2 General Concomitant Medications and Supportive Care Guidelines

Patients should be off any prior treatment or line of therapy at least 2 weeks prior

to D1 of induction therapy with the exception of hydrea. Hydrea will be allowed at the

discretion of the treating physician but must be stopped prior to starting CPX-351.

Necessary supportive measures for optimal medical care will be given throughout

the treatment as determined by the treating physician and the patient's medical needs. No

concomitant chemotherapy, immunotherapy, or therapy with monoclonal antibodies will

be allowed during the study.

Prophylactic antibiotics and antiviral agents (e.g. levofloxacin, valacyclovir, etc.)

are recommended while on study; however, the use of these or other drugs will be left to

the treating physician's discretion. Use of colony-stimulating factors or combinations

CASE 2918

Protocol Version 5.0

18 January 2021


thereof (e.g. G-CSF, GM-CSF, or erythropoietin) are at the discretion of the treating physician and are permitted if judged in the patient's best medical interest. At the D35 (+/- 10 days) bone marrow, if there is no evidence of blasts > 5%, G-CSF will be allowed to improve counts at the discretion of the treating physician.

## 6.3 Criteria for Removal from Study

In the absence of treatment delays due to adverse events, treatment may continue for one cycle of induction therapy and up to four cycles of consolidation therapy if patients achieve response criteria per section 12.0 or until one of the following criteria applies:

## End of Treatment Criteria:

- Disease progression (section 12.0),
- Intercurrent illness that prevents further administration of treatment,
- The investigator and/or treating physician considers it, for safety reasons, to be in the best interest of the subject. Unacceptable adverse events defined as following:
  - Any unacceptable treatment related grade 3 or 4 toxicities that fail to recover to baseline or < Grade 3 in the absence of treatment within 4 weeks
  - Impaired cardiac function
  - Severe OR life-threatening hypersensitivity reactions
  - Grade 4 non-hematological organ toxicities regardless of time to recovery, excluding:
    - Grade 4 fatigue, asthenia fever, anorexia or constipation
    - Grade 4 nausea, vomiting or diarrhea not requiring tube feeding, total parenteral nutrition, or requiring or prolonging hospitalization
    - Infection, bleeding, or other expected direct complication of cytopenias due to active underlying leukemia
    - Grade 4 infusion reaction including cytokine release syndrome (CRS), if successfully managed and which resolves within 72 hours
    - Grade 4 tumor lysis syndrome (TLS) if it is successfully managed clinically and resolves within 7 days without end-organ damage
    - Grade 4 isolated electrolyte abnormalities that last <72 hours
- Patient decision to withdraw from treatment (partial consent) or from the study (full consent),
- Pregnancy during the course of the study for a child-bearing participant
- Death while patient is on the study

Table 1: End of Treatment Criteria

## End of Study Criteria:

- Patient decision to withdraw from the study (full consent),
- Non-compliance with the study protocol,
- Death while patient is in the follow-up phase,
- Patient completed treatment and follow-up phase per protocol.

Table 2: End of Study Criteria

## 6.4 **Duration of Follow Up**

Following completion of active treatment (EOT) and while still on study (Follow up), patients will be followed for survival as for 1 year. During the first 6 months of follow-up, the patient will be seen in clinic as standard of care every 30 days, per the study calendar (section 11.2). The clinical course of all grade 3 or 4 events will be followed until resolution, stabilization, or until it has been determined study treatment or study participation is not the cause. New onset adverse events will not be recorded during follow-up.

Serious adverse events that are ongoing at the end of active treatment (EOT), will necessitate follow-up to determine the final outcome. Any serious adverse events that occur after the study period (EOT) and are considered related or possibly related to study treatment or study participation will be recorded and reported immediately, per institutional review board (IRB) requirement.

## 7.0 Dose Delays/Dose Modifications

No dose reductions of CPX-351 will be allowed during the study. Dose delays will be at the discretion of the treating physician after discussion with the PI. Missed doses of CPX-351 can be made up on subsequent days if felt to be in the best interest of the patient. CPX-351 doses must be given at least 24 hours apart. This will be determined by the treating physician following discussion with the PI.

If at any time during an infusion the patient experiences moderate hypersensitivity reactions, discontinuation of that infusion is mandatory. Premedicate with antihistamines and/or corticosteroids prior to all subsequent infusions. If a patient experiences a mild hypersensitivity reaction, regardless or premedication, infusion must be interrupted and can be re-initiated at half the prior rate.

#### 8.0 Adverse Events and Potential Risks

#### 8.1 Definitions

#### **8.1.1** Adverse Event

An **adverse event** (AE) is any unfavorable or unintended event, physical or psychological, associated with a research study, which causes harm or injury to a research participant as a result of the participant's involvement in a research study. The event can include abnormal laboratory findings, symptoms, or disease associated with the research study. The event does not necessarily have to have a causal relationship with the research, any risk associated with the research, the research intervention, or the research assessments.

Adverse events may be the result of the interventions and interactions used in the research; the collection of identifiable private information in the research; an underlying disease, disorder, or condition of the subject; and/or other circumstances unrelated to the research or any underlying disease, disorder, or condition of the subject.

#### **8.1.2** Serious Adverse Events

A **serious adverse event** (SAE) is any adverse experience occurring at any dose that results in any of the following outcomes:

- Results in death.
- Is a **life-threatening** adverse experience. The term life-threatening in the definition of serious refers to an adverse event in which the subject was at risk of death at the time of the event. It does not refer to an adverse event which hypothetically might have caused death if it were more severe.
- Requires inpatient hospitalization or prolongation of existing hospitalization. Any adverse event leading to hospitalization or prolongation of hospitalization will be considered as Serious, UNLESS at least one of the following expectations is met:
  - The admission results in a hospital stay of less than 24 hours OR

- The admission is pre-planned (e.g., elective or scheduled surgery arranged prior to the start of the study) OR
- The admission is not associated with an adverse event (e.g., social hospitalization for purposes of respite care.

However, it should be noted that invasive treatment during any hospitalization may fulfill the criteria of "medically important" and as such may be reportable as a serious adverse event dependent on clinical judgment. In addition, where local regulatory authorities specifically require a more stringent definition, the local regulation takes precedent.

- Results in persistent or significant disability/incapacity. The definition of disability is a substantial disruption of a person's ability to conduct normal life's functions.
- Is a congenital anomaly/birth defect.
- Is an **important medical event**. Important medical events that may not result death, be life-threatening, or require hospitalization may be considered a serious adverse experience when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood disease or disorders, or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse. The development of a new cancer is always considered an important medical event.

## **8.1.3** Adverse Event Evaluation

The investigator or designee is responsible for ensuring that all adverse events (both serious and non-serious) observed by the clinical team or reported by the subject which occur after the subject has signed the informed consent are fully recorded in the

subject's medical records. Source documentation must be available to support all adverse

events.

A laboratory test abnormality considered clinically relevant as deemed by the

treating physician should be reported as an adverse event.

The investigator or sub-investigator (treating physician if applicable) will provide

the following for all adverse events (both serious and non-serious):

• Event term (as per CTCAE)

• Description of the event

Date of onset and resolution

• Expectedness of the toxicity

Grade of toxicity

• Attribution of relatedness to the investigational agent- (this must be assigned

by an investigator, sub-investigator, or treating physician)

• Action taken as a result of the event, including but not limited to; no changes,

dose interrupted, reduced, discontinued, etc. or action taken with regard to the

event, i.e. no action, received conmed or other intervention, etc.

• Outcome of event

Descriptions and grading scales found in the NCI Common Terminology Criteria for

Adverse Events (CTCAE) version **5.0** will be utilized for AE reporting.


An expected adverse event is an event previously known or anticipated to result from

participation in the research study or any underlying disease, disorder, or condition of the

subject. The event is usually listed in the Investigator Brochure, consent form or research

protocol.

An unexpected adverse event is an adverse event not previously known or anticipated to

result from the research study or any underlying disease, disorder, or condition of the

subject.

CASE 2918 Protocol Version 5.0 **Attribution** is the relationship between an adverse event or serious adverse event and the study drug. Attribution will be assigned as follows:

- Definite The AE is clearly related to the study drug.
- Probable The AE is <u>likely related</u> to the study drug.
- Possible The AE <u>may be related</u> to the study drug.
- Unlikely The AE is <u>doubtfully related</u> to the study drug.
- Unrelated The AE is clearly NOT related to the study drug.

Protocol must specify if attribution is required for individual components of the treatment regimen or the treatment regimen as a whole.

## 8.2 Potential Risks of **CPX-351**

## COMMON, SOME MAY BE SERIOUS

In 100 people receiving CPX-351 more than 10 and up to 100 may have:

- Abdominal pain
- Anemia
- Anxiety
- Arrhythmia
- Chest pain
- Chills
- Constipation
- Cough
- Decreased appetite
- Delirium
- Diarrhea
- Dizziness
- Dyspnea
- Edema
- Fatigue
- Febrile neutropenia
- Fungal infection
- Headache
- Hemorrhage
- Hypertension
- Hypotension
- Hypoxia
- Rash
- Mucositis
- Musculoskeletal pain

- Nausea
- Neutropenia
- Non-conduction cardio toxicity
- Pleural effusion
- Pneumonia
- Pruritus
- Pyrexia
- Rash
- Sleep disorders
- Vomiting

## OCCASIONAL, SOME MAY BE SERIOUS

## In 100 people receiving CPX-351 from 4 to 20 may have:

- Acute renal failure
- Cellulitis
- Catheter/injection site reaction
- Ejection fraction decreased
- Fatigue
- Hemorrhoids
- Hypokalemia
- Malignant neoplasm progressive
- Petechiae
- Pneumonia
- Pyrexia
- Rash
- Sepsis
- Urinary tract infection
- Renal insufficiency
- Respiratory failure
- Transfusion reactions
- Upper respiratory induction (excluding fungal)
- Visual impairments (except bleeding)

## 8.3 SAE Report Form

SAEs will be recorded on the FDA Form 3500A (MedWatch) but should only be reported as instructed below. The electronic FDA SAE reporting forms should not be used.

## **8.4** Reporting Procedures for Serious Adverse Events

For the purposes of safety reporting, all adverse events will be reported that occur through 30 days after the final dose of study drug. Adverse events, both serious and non-

CASE 2918 Protocol Version 5.0 18 January 2021 serious, and deaths that occur during this period will be recorded in the source documents. All SAEs should be monitored until they are resolved or are clearly determined to be due to a subject's stable or chronic condition or intercurrent illness(es). Related AEs will be followed until resolution to baseline or grade 1 or stabilization.

## **8.4.1 SAE** Reporting Requirements

- Participating investigators (all sites) must report all serious adverse events to the
  Lead Site Principal Investigator (e.g. Sponsor-Investigator) within 24 hours of
  discovery or notification of the event. The participating investigator must also
  provide follow-up information on the SAE until final resolution.
- The Lead Site Principal Investigator will review the SAE and report the event to the FDA, external collaborator(s), and IRB as applicable.
- The Principal Investigator must send all SAEs (initial and follow-up) that require collection and reporting per protocol, and which occur in a subject who received CPX-351 as study drug, to Jazz Pharmaceuticals within 1 business day of their awareness of the SAE to AEreporting@jazzpharma.com.
- It is the Sponsor-Investigator's responsibility (e.g. lead site PI) to ensure that ALL serious adverse events that occur on the study (e.g. ALL SAEs that occur at each enrolling institution) are reported to all participating sites.

## **Institutional Review Board Reporting Requirements:**

• Investigative sites will report adverse events to their respective IRB according to the local IRB's policies and procedures in reporting adverse events.

## 8.5 SAEs and OnCore

- All SAEs will be entered into OnCore.
- A copy of the SAE form(s) submitted to the sponsor-investigator is also uploaded into Oncore.

## **8.6** Data Safety and Toxicity Committee

It is the responsibility of each site PI to ensure that ALL SAEs occurring on this trial (internal or external) are reported to the Case Comprehensive Cancer Center's Data

and Safety Toxicity Committee. This submission is simultaneous with their submission to

the sponsor and/or other regulatory bodies.

The sponsor-investigator is responsible for submitting an annual report to the

DSTC as per CCCC Data and Safety Monitoring Plan.

8.7 Data and Safety Monitoring Plan (DSMP)

This protocol will adhere to the policies of the Case Comprehensive Cancer

Center Data and Safety Monitoring Plan in accordance with NCI guidelines.

9.0 PHARMACEUTICAL INFORMATION

A list of the adverse events and potential risks associated with the investigational

or commercial agents administered in this study can be found in Section 8.

9.1 Investigational Agents

**9.1.1** Name of Agent

CPX-351

Other Names:

CPX-351

**Product description:** CPX-351 (daunorubicin and cytarabine) liposome for injection is a

combination of daunorubicin and cytarabine in a 1:5 molar ratio encapsulated in

liposomes for intravenous administration. The liposome membrane is composed of

distearoylphosphatidylcholine (DSPC), distearoylphosphatidylglycerol (DSPG), and

cholesterol in a 7:2:1 molar ratio.

**Solution preparation:** The appropriate number of vials of CPX-351

(cytarabine:daunorubicin) Liposome Injection should be removed from the refrigerator

prior to reconstitution. Reconstitute with 19 mL of sterile water for injection using a 20

mL syringe. Do not heat CPX-351 (cytarabine:daunorubicin) Liposome Injection. After

reconstitution, invert vials gently 3-4 times and let rest for 15 minutes and repeat vial

inversion prior to withdrawing drug for dilution. The concentration of the reconstituted

dispersion is 5 mg-2.2mg/mL (cytarabine-daunorubicin). CPX-351 should be diluted in

approximately 500 mL of sodium chloride injection or dextrose injection.

The IV bags and infusion sets must be non-DEHP. Aseptic technique must be strictly

observed throughout the handling of CPX-351 (cytarabine:daunorubicin) Liposome

CASE 2918 Protocol Version 5.0


Injection since no bacteriostatic agent or preservative is present. The infusion of CPX-351 (cytarabine:daunorubicin) Liposome Injection must be started within 4 hours of dilution. Vials are for single use. Unused material should be recorded as such and discarded according to institutional policies. Procedures for proper handling and disposal of anticancer drugs should be implemented.

**Storage requirements:** Store un-reconstituted CPX-351 vials in a refrigerator at 2°C to 8°C (36°F to 46°F) in an upright position. The vial should be stored in its original carton to protect from light.

**Stability:** If the diluted infusion solution is not used immediately, store in refrigerator at 2°C to 8°C for up to 4 hours.

Route of administration: The infusion of CPX-351 (cytarabine:daunorubicin) Liposome Injection will be performed through a central venous catheter, using an infusion pump to ensure that the drug is infused over the specified time period. Non-DEHP containing administration sets should be used. **Do not use an in-line filter.** CPX-351 should never be given by the intramuscular or subcutaneous route. Administer CPX-351 over approximately 90 minutes via an infusion pump. Flush the line to ensure administration of the full dose. The dosage (total mg/m²), start/stop time of the infusion, total volume infused, must be documented in the patient's chart.

**<u>Drug Procurement:</u>** CPX-351 will be supplied for this study by Jazz Pharmaceutical.

**Drug Accountability:** The study pharmacist or designee must maintain records of the delivery of CPX-351 to the study site, the inventory at the site, the use by each patient, and the disposition of unused product. These records should include dates, quantities, lot numbers, expiration dates and patient identifications. Institutions should maintain records that document adequately that the patients were provided the doses specified by the protocol and reconcile all investigational product received from the Sponsor. Records of storage conditions (temperature logs) must be kept for the entire period that CPX-351 is maintained at the institution.

**<u>Drug Destruction</u>**: At the completion of the study, there will be a final reconciliation of drug shipped, drug consumed, and drug remaining. This reconciliation will be logged on

CASE 2918 Protocol Version 5.0 the drug reconciliation form, signed and dated. Any discrepancies noted will be investigated, resolved, and documented prior to return or destruction of unused study drug. Drug destroyed on site will be documented in the study files.

## 10.0 EXPLORATORY or CORRELATIVE STUDIES

Bio specimens (whole blood, 10 mL) will be collected as outlined in section 11.2 at screening, C1D35 (+/- 10 days) and EOT for general research purposes, potentially including genetic analysis research. All subjects must consent to provide archived sample for future research.

All samples obtained will be stored at the Cleveland Clinic Translational Hematology and Oncology Research laboratory. Samples will remain at the Cleveland Clinic to be used for research purposes for this study as well as for future research projects approved by the IRB.

## **10.1 Collection of Samples**

10mL of whole blood will be collected in an extra lab tube at screening, C1D35 (+/- 10 days) and EOT (section 11.2). Details and instructions about the collection, processing and shipping can be found in the Lab Manual. All samples will be housed at and should be delivered and/or shipped to:

Principle Research Technologists
Translational Hematology and Oncology Laboratory
Cleveland Clinic, LC – NE6 – 250
9620 Carnegie, Avenue
Cleveland, OH 44195
Phone: (216) 444-0256

## 11.0 STUDY PARAMETERS AND CALENDAR

## 11.1 Study Parameters

- 11.1.1 Screening Evaluations (Consent to D-1)
  - 1. History and physical examination.
  - 2. ECOG performance status (Appendix I).

CASE 2918 Protocol Version 5.0 18 January 2021

- 3. Vitals.
- 4. Hematology exam (Appendix IV).
- 5. Serum chemistry exam (Appendix IV).
- 6. Echocardiogram and electrocardiogram (If completed prior to consent and within 28 days of C1D1, may count towards screening procedures).
- 7. Bone marrow aspirate and biopsy, including cytogenetics, within 28 days of therapy start to confirm diagnosis (If completed prior to consent and within 28 days of C1D1, may count towards screening procedures).
- 8. Serum pregnancy test for women of childbearing potential within Child bearing potential is defined as not post-menopausal for 12 months or no previous surgical sterilization.
- 9. Documentation in the medical record (consisting of start date, dose, frequency, route, and if applicable stop date) of all medications including vitamins and other over the counter medications.
- 10. Documentation in the medical record (consisting of start and stop date, dose, frequency and route) of any prior administration of cancer agent therapy.
- 11. Documentation in the medical record of all adverse events (graded per CTCAE V.5.0) present at baseline. Documentation must include start and stop dates (if resolved), relationship to CPX-351 and grade.
- 11.1.2 Induction Therapy (C1D1 to C1D35 and/or count recovery).
  - 1. Physical examination will occur daily while inpatient (Appendix IV).
  - 2. ECOG performance status will be collected daily while in-patient (Appendix I).
  - 3. Vitals will be collected daily while in-patient (Appendix IV).
  - 4. Echocardiogram will be completed on day 1 prior to dosing.
  - 5. Hematology exam on days 1-5, and twice weekly during days 6-27 (Appendix IV).
  - 6. Serum chemistry exam on days 1-5, and twice weekly days 6-27 (Appendix IV).
  - 7. Administration of CPX-351 at  $44 \text{mg/m}^2$  on days 1, 3 and 5.
  - 8. Bone marrow aspirate and biopsy, including cytogenetics, on D35 (+/- 10 days)

- 9. Disease response assessment will be assessed by the treating physician on D35 (+/- 10 days) (Table 2).
- 10. Serum pregnancy test on C1D1 only for women of childbearing potential. Child bearing potential is defined as not post-menopausal for 12 months or no previous surgical sterilization.
- 11. Documentation in the medical record (consisting of start date, dose, frequency, route, and if applicable stop date) of all medications including vitamins and other over the counter medications.
- 12. Documentation in the medical record (consisting of start and stop date, dose, frequency and route) of any prior administration of cancer agent therapy.
- 13. Documentation in the medical record of all adverse events (graded per CTCAE V.5.0). Documentation must include start and stop dates (if resolved), relationship to CPX-351 and grade.

## Consolidation Therapy (C2D1 to C5D28)

- 1. Physical examination on day 1 of each 28 day cycle (Appendix IV).
- 2. ECOG performance status will be collected on day 1 of each 28 day cycle (Appendix I).
- 3. Vitals will be collected prior to dosing on days 1 and 3 (Appendix IV).
- 4. Echocardiogram will be completed prior to dosing on day 1 of every cycle
- 5. Hematology exam on dosing days 1 and 3 of and twice weekly during each 28 day cycle (Appendix IV).
- 6. Serum chemistry exam on dosing days 1 and 3 and twice weekly during each 28 day cycle (Appendix IV).
- 7. Administration of CPX-351 at 15.4mg/m² (daunorubicin 15.4 mg/m² and cytarabine 35 mg/m²) on days 1 and 3 of every 28 day cycle
- 8. Serum pregnancy test will be collected on day 1 of every 28 day cycle, only for women of childbearing potential. Child bearing potential is defined as not postmenopausal for 12 months or no previous surgical sterilization.

- 9. Documentation in the medical record (consisting of start date, dose, frequency, route, and if applicable stop date) of all medications including vitamins and other over the counter medications will be collected on day one of every 28 day cycle.
- 10. Documentation in the medical record (consisting of start and stop date, dose, frequency and route) of any prior administration of cancer agent therapy will be collected on day one of every 28 day cycle.
- 11. Documentation in the medical record of all adverse events (graded per CTCAE V.5.0). Documentation must include start and stop dates (if resolved), relationship to CPX-351 and grade will be collected on day one of every 28 day cycle.

## End of Treatment (EOT)

- 1. Physical examination (Appendix IV).
- 2. ECOG performance status (Appendix I).
- 3. Vitals (Appendix IV).
- 4. Hematology exam (Appendix IV).
- 5. Serum chemistry exam (Appendix IV).
- 6. Bone marrow aspirate and biopsy, including cytogenetics.
- 7. Disease assessment (Table 2).
- 8. Documentation in the medical record (consisting of start date, dose, frequency, route, and if applicable stop date) of all medications including vitamins and other over the counter medications will be collected.
- Documentation in the medical record (consisting of start and stop date, dose, frequency and route) of any prior administration of cancer agent therapy will be collected.
- 10. Documentation in the medical record of all adverse events (graded per CTCAE V.5.0). Documentation must include start and stop dates (if resolved), relationship to CPX-351 and grade will be collected.

# 11.2 Calendar

| | | | | | | | | | | | | | т т | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | Screening<br>Period | | Indu | iction ] | | e<br>cycle | | | Consolidation Phase Up to 4 cycles | | | | End of<br>Treatment<br>(EOT) | Follow-<br>up <sup>g</sup> |
| Day | 28 Days | 1 | 2 | 3 | 4 | 5 | 6-27 | 35 <sup>1</sup> | 1 <sup>dij</sup> | $\frac{2}{2}$ | 3 | 4 - 28 | | |
| CPX-351 Administration <sup>a</sup> | | X | | X | | X | | | X | | X | | | |
| Informed Consent Form (ICF) | X | | | | | | | | | | | | | |
| Disease history and prior therapies | X | | | | | | | | | | | | | |
| History and physical exam <sup>b</sup> | X | | | | | | | | X | | | | X | |
| Vital signs <sup>b</sup> | X | Xop | | Xop | | | | X | Xop | | Xop | | | |
| Concomitant medications | X | X | | | | | | | X | | | | X | |
| ECOG performance status <sup>c</sup> | X | | | | | | | | X | | | | X | |
| Hematology <sup>b</sup> | X | X | X | X | X | X | X <sup>n</sup> | X | Xe | | | X <sup>n</sup> | X | $X^g$ |
| Serum chemistry <sup>b</sup> | X | X | X | X | X | X | Xn | X | Xe | | | X <sup>n</sup> | X | |
| Pregnancy test | X | X <sup>k</sup> | | | | | | | X <sup>k</sup> | | | | | |
| Echocardiogram | Xr | Xq | | | | | | | X | | | | | |
| Electrocardiogram | Xr | | | | | | | | | | | | | |
| Bone marrow biopsy and aspiration <sup>b</sup> | Xr | | | | | | | X | | | | | X | |
| Disease response assessment <sup>f</sup> | X | | | | | | | X | | | | | X | |
| Correlative analysis blood draw <sup>m</sup> | X | | | | | | | X | | | | | X | |
| Survival follow-up | | | | | | | | | | | | | | $X^h$ |
| Adverse event assessment | | | | | | | <del>(</del> | $X \rightarrow$ | | _ | | | | |

- a: During the induction phase all patients will receive 44mg/m<sup>2</sup>. Following the induction phase if patients achieve a response (per section 12.0) they may continue onto the consolidation phase. During the consolidation phase patients will receive 15.4mg/m<sup>2</sup> (daunorubicin 15.4 mg/m<sup>2</sup> and cytarabine 35 mg/m<sup>2</sup>) for up to 4 cycles.
- b: See Appendix IV for required tests.
- c: See Appendix I for performance status grading.
- d: Indicates at +/-3 day window.
- e: Required twice weekly to monitor counts, can be completed at a local laboratory.
- f: See Section 12.0 for MDS response assessment criteria.
- g: Follow up will occur monthly as SOC for the first 6 months of follow-up. See section 6.4 for adverse event reporting requirements.
- h: Survival Follow up will occur bimonthly (60 days) for a duration of 1 year from patient's EOT visit.
- i: During only the first cycle in consolidation phase, CPX-351 must be given no earlier than 35 days after the start of induction and no later than 75 days after the start of induction. There should be 35 days between the start of each subsequent consolidation cycles Patients must have recovered to ANC >500/µL and platelets >50,000/µL to be eligible for any consolidation therapy.
- j: Prior to the first cycle of consolidation therapy, patient must have an ECOG PS of 0-2.
- k: Must be negative prior to dosing.
- 1: Indicates a +/-10 day window.
- m: 10mL of whole blood will be collected in an extra lab tube for these tests.
- n: Hematology and serum chemistry will be assessed 1-3x weekly at the discretion of the treating physician to monitor counts. These can be completed at a local laboratory.
- o: On dosing days, for induction phase only, vitals must be collected prior to infusion, 5, 10, 30 and 60 minutes post the start of infusion and at the end of infusion. On dosing days, for consolidation phase, vitals must be collected prior to infusion and at the end of infusion.
- p: Indicates a (+/-) 5 minute window.
- q: Required if patient has not had an ECHO within 28 days of C1D1.
- r: If completed prior to consent and within 28 days of C1D1, may count towards screening procedures.
## 12.0 MEASUREMENT OF EFFECT

Response criteria will be defined by the IWG criteria ET 2006. Patients will be assessed for response at the end of induction cycle.

Response criteria will be defined as follow:

| Response | Definition |
|---|---|
| | Responses must be for at least 4 weeks) |
| Complete remission | Marrow: |
| (CR) | < 5% myeloblasts with normal maturation |
| | of all cell lines. |
| | Persistent dysplasia will be noted (dysplastic |
| | changes should consider the normal range of |
| | dysplastic changes.) |
| | Blood: |
| | - Hemoglobin (Hgb) $\geq$ 11 g/dL (un |
| | transfused, patient not on EPO) |
| | - Neutrophils $\geq 1 \times 109 / L$ (not on myeloid |
| | growth factor) |
| | - Platelets $\geq 100 \times 109/L$ (not on |
| | thrombopoietic agent) |
| | - No blasts |
| Partial remission (PR) | All CR criteria (if abnormal prior to |
| | treatment), except: |
| | Marrow blasts decreased by ≥50% |
| | compared with pretreatment but still > 5%. |
| M CD | Cellularity and morphology not relevant |
| Marrow CR | Marrow: |
| | $\leq$ 5% myeloblasts and decrease by $\geq$ 50% |
| | over pretreatment Blood: |
| | if hematologic improvement (HI) responses, they will be noted in |
| | addition to the marrow CR |
| Stable disease (SD) | Failure to achieve at least PR, but no |
| State disease (SD) | evidence of progression for > 8 weeks |
| Failure | Death during treatment or disease |
| 1 411410 | progression characterized by worsening of |
| | cytopenias, increase in percentage of |
| | marrow blasts, or progression to an MDS |
| | FAB subtype more advanced than |
| | pretreatment. |
| | l Production. |

| Relapse after CR or PR (PD) | At least one of the following: - Return to pretreatment bone marrow blast percentage - Decrement of ≥ 50% from maximum remission/response levels in granulocytes or platelets - Reduction in Hgb concentration by ≥ 1.5 g/dL or transfusion dependence (in the absence of another explanation, such as acute infection, GI bleeding, hemolysis, etc.) |
|---|---|
| Cytogenetic response | Complete: Disappearance of the chromosomal abnormality without appearance of new ones Partial: At least 50% reduction of the chromosomal abnormality |
| Hematologic Improvement | Response Criteria |
| D 4 11 | (responses must last at least 8 weeks) |
| Erythroid response | Hgb increase by $\geq 1.g/dL$ |
| (pretreatment, $< 11 \text{ g/dL}$ ) | Relevant reduction of units of RBC |
| | transfusions by an absolute number of at |
| | least 4 RBC transfusions/8wk compared |
| | with the pretreatment transfusion number in |
| | the previous 8 wk. |
| | Only RBC transfusions given for a Hgb of ≤ |
| | 9 g/dL pretreatment will count in the RBC |
| D1 . 1 . | transfusion response evaluation |
| Platelet response | Absolute increase of $\geq 30 \times 109/L$ for |
| (pretreatment, $< 100 \times 109 / L$ ) | patients starting with > 20 x<br>109/L |
| | Increase from $< 20 \times 109/L$ to $> 20 \times 109/L$ |
| | and by at least 100% |
| Neutrophil response | At least 100% increase an absolute increase |
| (pretreatment, $< 1 \times 109/L$ ) | > 0.5 x 109/L |
| Progression or relapse after HI | At least 1 of the following: |
| | At least 50% decrement from maximum |
| | response levels in granulocyte or platelets |
| | Reduction in Hgb by $\geq 1.5$ g/dL |
| | J J = - 0 |
| | Transfusion dependence (in the absence of |
| | Transfusion dependence (in the absence of another explanation, such as acute infection, |

Table 3: Response Criteria for MDS Patients

13.0 **DATA REPORTING / REGULATORY CONSIDERATIONS** 

Adverse event lists, guidelines, and instructions for AE reporting can be found in Section

8.0 (Adverse Events: List and Reporting Requirements).

13.1 **Data Reporting** 

The OnCore® Database will be utilized, as required by the Case Comprehensive

Cancer Center, to provide data collection for both accrual entry and trial data

management. OnCore® is a Clinical Trials Management System housed on secure

servers maintained at Case Western Reserve University. OnCore® Access to data

through OnCore® is restricted by user accounts and assigned roles. Once logged into the

OnCore® system with a user ID and password, OnCore® defines roles for each user

which limits access to appropriate data. User information and password can be obtained

by contacting the OnCore® Administrator at OnCore-registration@case.edu.

OnCore® is designed with the capability for study setup, activation, tracking,

reporting, data monitoring and review, and eligibility verification. This study will utilize

electronic Case Report Form completion in the OnCore® database. A calendar of events

and required forms are available in OnCore®.

13.2 **Regulatory Considerations** 

The study will be conducted in compliance with ICH guidelines and with all

applicable federal (including 21 CFR parts 56 & 50), state or local laws.


13.2.1 Written Informed consent

Provision of written informed consent must be obtained prior to any study-related

procedures. The Principal Investigator will ensure that the subject is given full and

adequate oral and written information about the nature, purpose, possible risks and

benefits of the study as well as the subject's financial responsibility. Subjects must also

be notified that they are free to discontinue from the study at any time. The subject

**CASE 2918** Protocol Version 5.0 should be given the opportunity to ask questions and be allowed time to consider the

information provided.

The original, signed written Informed Consent Form must be kept with the

Research Chart in conformance with the institution's standard operating procedures. A

copy of the signed written Informed Consent Form must be given to the subject.

Additionally, documentation of the consenting process should be located in the research

chart.

13.2.2 Subject Data Protection

In accordance with the Health Information Portability and Accountability Act

(HIPAA), a subject must sign an authorization to release medical information to the

sponsor and/or allow the sponsor, a regulatory authority, or Institutional Review Board

access to subject's medical information that includes all hospital records relevant to the

study, including subjects' medical history.

13.2.3 Retention of records

The Principal Investigator of The Case Comprehensive Cancer Center supervises

the retention of all documentation of adverse events, records of study drug receipt and

dispensation, and all IRB correspondence for as long as needed to comply with local,

national and international regulations. No records will be destroyed until the Principal

Investigator confirms destruction is permitted.

13.2.4 Audits and inspections

Authorized representatives of the sponsor, a regulatory authority, an Independent

Ethics Committee (IEC) or an Institutional Review Board (IRB) may visit the site to

perform audits or inspections, including source data verification. The purpose of an audit

or inspection is to systematically and independently examine all study-related activities

and documents to determine whether these activities were conducted, and data were

recorded, analysed, and accurately reported according to the protocol, Good Clinical

Practice (GCP), guidelines of the International Conference on Harmonization (ICH), and


**CASE 2918** Protocol Version 5.0

any applicable regulatory requirements. For multi-center studies, participating sites must inform the sponsor-investigator of pending audits.

#### 14.0 STATISTICAL CONSIDERATIONS

In determining the sample size for the patient cohort, Minimax Simon's two-stage design (Simon, 1989) will be used. The null hypothesis that the true response rate is 0.1 will be tested against a one sided alternative. In the first stage, 7 patients will be accrued in each arm. If there are two or less responses in these 7 patients, the arm will be stopped. Interim analysis will conducted to determine the benefit of applying the drug in each arm. In the winning arm, 11 additional patients will be accrued for a total of 18. The null hypothesis will be rejected if 4 or more responses are observed in 18 patients. This design yields a type I error rate of 0.1 and power of 0.8 when the true response rate is 0.3.

Descriptive statistical analysis will be calculated, including histograms or boxplots, proportions, range, means and standard deviations. Fisher's exact test and Wilcoxon rank test will be used in univariate analyses of categorical and continuous variables, respectively. Overall response (CR + CRi +) rate and its 95% CI. Given there is no adjustment for multiple comparisons, need to note the p-values from the univariate analyses will be nominal and not used to infer significance.

#### **Toxicity Monitoring Rules**

The following toxicity monitoring plan will terminate the trial early given evidence for excessive rates of toxicity with CPX-351based on the method of Thall et al.  $^{14}$  Early termination will be applied to evaluate patients experiencing toxicity defined as any grade  $\geq 3$  non-hematologic AE that is determined to be at least possibility related to CPX-351. A total of 25 patients will be enrolled. The monitoring rules target a toxicity rate of 20% and assume a non-informative Beta (0.2, 0.8) prior distribution. The trial will stop early for toxicity if Pr(Toxicity Rate  $> 0.20 \mid data) > 0.85$ , i.e. stop early if the evidence for excessive toxicity (higher than 20%) for the target population given observed data is sufficiently high (probability > 0.85). Monitoring will be carried out

from the 3rd patient. Table 5 summarizes the resultant stopping boundaries and Table 6 summarizes the trial's operating characteristics.

Table 5. Summary of early stopping boundaries from the 3rd patient. Target toxicity rate is 20%. Using prior of Beta (0.2, 0.8) and posterior probability threshold of 0.85. E.g. If 3 or more patients experience grade  $\geq 3$  non-hematologic AEs out of the first 6 patients, the trial will stop early. Whenever a grade  $\geq 3$  non-hematologic AE is observed, check this table to see if the boundary has been crossed. E.g. if a total of 4 grade  $\geq 3$  non-hematologic AEs has been observed on trial, and the total number of patients treated is 9 or less, then stop the trial for excessive toxicity.

| Stop Early if #Patients Experienced grade | | 3 | 4 | 5 | 5 | 6 | 7 | 8 |
|---|---|---|---|---|---|---|---|---|
| ≥3 non-hematologic AE | | | | | | | | |
| Total #Patients Treated | 3 | 6 | 9 | 12 | 15 | 18 | 21 | 24 |

Table 6. Summary of operating characteristics based on 10,000 simulations using boundaries in Table 5 for early stopping. For example, if the true toxicity rate is 20%, the probability of early stopping is 0.27, and if the true toxicity rate is 40%, the probability of early stopping is 0.88.

| Scenario | True Toxicity | Pr(Early | Average #Patients | Average |
|----------|---------------|----------|-------------------|-------------|
| | Rate | Stop) | Treated | #Toxicities |
| 1 | - 0.10 | 0.05 | 23.2 | 2.3 |
| 2 | 0.20 | 0.27 | 19.8 | 4.0 |
| 3 | 0.30 | 0.62 | 14.6 | 4.4 |
| 4 | 0.40 | 0.88 | 9.8 | 3.9 |

Summary statistics of toxicity will be provided in frequencies and percentages.

Toxicity rate will be estimated along with 95% CIs. Other statistical analyses will be carried out as appropriate.

#### REFERENCES

- 1. Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G *et al.* International scoring system for evaluating prognosis in myelodysplastic syndromes. *Blood* 1997; **89**(6): 2079-88.
- 2. Kantarjian H, O'Brien S, Ravandi F, Cortes J, Shan J, Bennett JM *et al.* Proposal for a new risk model in myelodysplastic syndrome that accounts for events not considered in the original International Prognostic Scoring System. *Cancer* 2008; **113**(6): 1351-61.
- 3. Malcovati L, Germing U, Kuendgen A, Della Porta MG, Pascutto C, Invernizzi R et al. Time-dependent prognostic scoring system for predicting survival and leukemic evolution in myelodysplastic syndromes. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology* 2007; **25**(23): 3503-10.
- 4. Nazha A, Komrokji RS, Garcia-Manero G, Barnard J, Roboz GJ, Steensma DP *et al.* The efficacy of current prognostic models in predicting outcome of patients with myelodysplastic syndromes at the time of hypomethylating agent failure. *Haematologica* 2016; **101**(6): e224-7.
- 5. Nazha A, Sekeres MA, Komrokji R, Steensma DP, Kantarjian H, Roboz G *et al.* Validation of a post-hypomethylating agent failure prognostic model in myelodysplastic syndromes patients treated in a randomized controlled phase III trial of rigosertib vs. best supportive care. *Blood cancer journal* 2017; 7(12): 644.
- 6. Prebet T, Fenaux P, Vey N. Predicting outcome of patients with myelodysplastic syndromes after failure of azacitidine: validation of the North American MDS consortium scoring system. *Haematologica* 2016; **101**(10): e427-e428.
- 7. Feldman EJ, Lancet JE, Kolitz JE, Ritchie EK, Roboz GJ, List AF *et al.* First-In-Man Study of CPX-351: A Liposomal Carrier Containing Cytarabine and Daunorubicin in a Fixed 5:1 Molar Ratio for the Treatment of Relapsed and Refractory Acute Myeloid Leukemia. *Journal of Clinical Oncology* 2011; **29**(8): 979-985.
- 8. Cortes JE, Goldberg SL, Feldman EJ, Rizzeri DA, Hogge DE, Larson M *et al.* Phase II, multicenter, randomized trial of CPX-351 (cytarabine:daunorubicin) liposome injection versus intensive salvage therapy in adults with first relapse AML. *Cancer* 2015; **121**(2): 234-42.
- 9. Lancet JE, Uy GL, Cortes JE, Newell LF, Lin TL, Ritchie EK *et al.* CPX-351 (cytarabine and daunorubicin) Liposome for Injection Versus Conventional Cytarabine Plus Daunorubicin in Older Patients With Newly Diagnosed

- Secondary Acute Myeloid Leukemia. *Journal of Clinical Oncology* 2018; **36**(26): 2684-2692.
- 10. Festuccia M, Baker K, Gooley TA, Sandmaier BM, Deeg HJ, Scott BL. Hematopoietic Cell Transplantation in Myelodysplastic Syndromes after Treatment with Hypomethylating Agents. *Biology of blood and marrow transplantation : journal of the American Society for Blood and Marrow Transplantation* 2017; **23**(9): 1509-1514.
- 11. Ball B, Komrokji RS, Ades L, Sekeres MA, DeZern AE, Pleyer L *et al*. Evaluation of induction chemotherapies after hypomethylating agent failure in myelodysplastic syndromes and acute myeloid leukemia. *Blood advances* 2018; **2**(16): 2063-2071.
- 12. Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM *et al.* The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. *Blood* 2016; **127**(20): 2391-405.
- 13. Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD *et al.* Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. *Blood* 2006; **108**(2): 419-25.

# APPENDIX I

#### PERFORMANCE STATUS CRITERIA

| EC | OG Performance Status Scale | Karnofsky Performance Scale | |
|---|---|---|---|
| Grade | Description | Percent | Description |
| Normal activity. Full active, able | | 100 | Normal, no complaints, no evidence of disease. |
| 0 | | | Able to carry on normal activity; minor signs or symptoms of disease. |
| | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able | 80 | Normal activity with effort; some signs or symptoms of disease. |
| 1 | to carry out work of a light or<br>sedentary nature (e.g., light<br>housework, office work). | 70 | Cares for self, unable to carry on normal activity or to do active work. |
| | In bed < 50% of the time. Ambulatory and capable of all | | Requires occasional assistance, but is able to care for most of his/her needs. |
| 2 | self-care, but unable to carry out any work activities. Up and about more than 50% if waking hours. | 50 | Requires considerable assistance and frequent medical care. |
| | In bed > 50% of the time. Capable of only limited self-care, | 40 | Disabled, requires special care and assistance. |
| 3 confined to bed or chair more than 50% of waking hours. | | 30 | Severely disabled,<br>hospitalization indicated.<br>Death not imminent. |
| | 100% bedridden. Completely disabled. Cannot carry on any | 20 | Very sick, hospitalization indicated. Death not imminent. |
| 4 | self-care. Totally confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. |
| 5 | Dead. | 0 | Dead |

## **APPENDIX II: STUDY DESIGN TIME POINT DEFINITIONS**

| Study Time Points | Definitions |
|---|---|
| Screening | The screening period will occur over 28 |
| | days from the time of consent to day -1. |
| Induction Period | Day 1 <sup>a</sup> to D35 and/or count recovery |
| Disease Response | The D35 (+/-10 days) bone marrow. |
| Consolidation Period | The consolidation period is defined as |
| | C2D1 through C5D28. Patients who meet |
| | disease response criteria will be eligible to |
| | receive up to 4 cycles of consolidation |
| | therapy. |
| End of Treatment (EOT) | The day patients meets the defined EOT |
| | criteria (Table 1) and discontinues study |
| | treatment. |
| Follow up | Patient will be followed monthly as SOC |
| | every 30 days for the duration of 6 months |
| | after EOT. |
| End of Study (EOS) | The time the patient completes 1 year of |
| | follow up and/or patient's death, whichever |
| | were to occur first. |
| a: Day 1 is defined as the first dose of CPX- | 351 |

## **APPENDIX IV: STUDY DESIGN TIME POINT DEFINITIONS**

| <u>Hematology</u> | <u>Serum</u> | <u>Vitals</u> | <u>Physical</u> | Bone Marrow Biopsy |
|---|---|---|---|---|
| | <u>Chemistry</u> | | <u>Exam</u> | <u>&amp; Aspirate</u> |
| RBC count | Total protein | Temperature | Height <sup>a</sup> | Marrow blast percent |
| WBC count | Albumin | Respirations | Weight <sup>b</sup> | Marrow cellularity |
| Hematocrit | Sodium | Blood Pressure | | Auer Rods |
| Hemoglobin | Potassium | Pulse | | Dysplasia |
| MCV | Chloride | | | Cytogenetics |
| MCHC | Bicarbonate | | | |
| Platelet count | Glucose | | | |
| Neutrophils | AST | | | |
| Eosinophils | ALT | | | |
| Basophils | Creatinine | | | |
| Monocytes | Calcium | | | |
| Lymphocytes | Bilirubin | | | |
| Blast percent | Alkaline | | | |
| | phosphate | | | |
| | Phosphorus | | | |
| | Uric acid | | | |
| | Magnesium | | | |
| a. IIaialet | ulry be sellested a | | | |

a: Height will only be collected at screeningb: On dosing days, weight will be collected prior to dosing

#### APPENDIX V: Post-HMA Failure Model



| Parameter at HMA failure | Score |
|---------------------------------------|-------|
| ECOG Performance status > 1 | 1.0 |
| Complex Karyotype (≥ 4 abnormalities) | 1.0 |
| Age, years | |
| > 75 - <u>&lt;</u> 84 | 1.0 |
| > 84 | 2.0 |
| Bone Marrow Blast > 20 % | .75 |
| Transfusion dependent (yes) | .75 |
| Platelets × 10 <sup>9</sup> /L | |
| < 30 | 1.0 |

# **Post-HMA Failure Model**

CASE 2918 Protocol Version 5.0 18 January 2021